CLINICAL TRIAL: NCT05501366
Title: Strategies to Augment Ketosis: Optimization of Ketone Delivery Strategies
Acronym: STAK: OK'd
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jeff Volek, Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2022H0160; CDMRP-PR212399-A (Other Grant/Funding Number: Departentof Defense)
Record Dates: First submitted 2022-08-01; First posted 2022-08-15 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Ketosis
MeSH Terms: conditions — Ketosis | interventions — Blood Specimen Collection; Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- BHB Mono-ester 180mg/kg (Experimental)
  Interventions: Dietary Supplement: Ketone Supplement; Behavioral: Beverage Tolerability Questionnaire (BTQ) and satiety visual analogue scale; Biological: Blood Draw; Other: Breath Reading; Other: Heart Rate Variability; Other: CGM/CKM; Other: Urine Analysis
- BHB mono-ester 360mg/kg (Experimental)
  Interventions: Dietary Supplement: Ketone Supplement; Behavioral: Beverage Tolerability Questionnaire (BTQ) and satiety visual analogue scale; Biological: Blood Draw; Other: Breath Reading; Other: Heart Rate Variability; Other: CGM/CKM; Other: Urine Analysis
- C8 Ketone Di-ester 180mg/kg (Experimental)
  Interventions: Dietary Supplement: Ketone Supplement; Behavioral: Beverage Tolerability Questionnaire (BTQ) and satiety visual analogue scale; Biological: Blood Draw; Other: Breath Reading; Other: Heart Rate Variability; Other: CGM/CKM; Other: Urine Analysis
- C8 Ketone Di-ester 360mg/kg (Experimental)
  Interventions: Dietary Supplement: Ketone Supplement; Behavioral: Beverage Tolerability Questionnaire (BTQ) and satiety visual analogue scale; Biological: Blood Draw; Other: Breath Reading; Other: Heart Rate Variability; Other: CGM/CKM; Other: Urine Analysis
- AcAc Di-ester 180mg/kg (Experimental)
  Interventions: Dietary Supplement: Ketone Supplement; Behavioral: Beverage Tolerability Questionnaire (BTQ) and satiety visual analogue scale; Biological: Blood Draw; Other: Breath Reading; Other: Heart Rate Variability; Other: CGM/CKM; Other: Urine Analysis
- AcAc Di-ester 360mg/kg (Experimental)
  Interventions: Dietary Supplement: Ketone Supplement; Behavioral: Beverage Tolerability Questionnaire (BTQ) and satiety visual analogue scale; Biological: Blood Draw; Other: Breath Reading; Other: Heart Rate Variability; Other: CGM/CKM; Other: Urine Analysis
- (R)-1,3 butanediol 180mg/kg (Experimental)
  Interventions: Dietary Supplement: Ketone Supplement; Behavioral: Beverage Tolerability Questionnaire (BTQ) and satiety visual analogue scale; Biological: Blood Draw; Other: Breath Reading; Other: Heart Rate Variability; Other: CGM/CKM; Other: Urine Analysis
- (R)-1,3 butanediol 360mg/kg (Experimental)
  Interventions: Dietary Supplement: Ketone Supplement; Behavioral: Beverage Tolerability Questionnaire (BTQ) and satiety visual analogue scale; Biological: Blood Draw; Other: Breath Reading; Other: Heart Rate Variability; Other: CGM/CKM; Other: Urine Analysis
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Ketone Supplement; Behavioral: Beverage Tolerability Questionnaire (BTQ) and satiety visual analogue scale; Biological: Blood Draw; Other: Breath Reading; Other: Heart Rate Variability; Other: CGM/CKM; Radiation: DXA; Other: Urine Analysis

INTERVENTIONS:
Dietary Supplement: Ketone Supplement — Four different exogenous ketone products at two serving sizes or a non-ketogenic placebo (one study product per test day). 1) Monoester of BHB (R)-1,3 butanediol (BHB Mono-ester), 2) diester of hexanoic acid (a ketogenic medium chain fatty acid) and (R)-1,3 butanediol (C6 Di-ester) 3) diester of AcAc and (R,S)-1,3 butanediol (AcAc Di-ester) & 4) (R) -1,3 butanediol only (BDO). All products will be delivered in 2 different dosages 180mg/kg and 360mg/kg on separate testing days.
Behavioral: Beverage Tolerability Questionnaire (BTQ) and satiety visual analogue scale — Beverage Tolerability Questionnaire (BTQ) and satiety visual analogue scale will be administered at beginning and end of testing day to tests palatability of supplement
Biological: Blood Draw — IV cannula will be inserted at the start of each Test Day, and removed at the end of each Test Day, Blood samples will be collected according to the schedule in Figure 1. Cannula will be flushed with a small volume of saline after each sample to maintain patency. We will draw 504 mL of blood, which is about 2.1 cups throughout the 4-week intervention
Other: Breath Reading — Participants will breathe into a commercially available handheld breath acetone analyzer according to the schedule. Participants will wear a fitted face mask attached to a metabolic cart for a 10-minute period every 60 minutes
Other: Heart Rate Variability — Participants will wear a Bluetooth heart rate monitor chest strap throughout the test day.
Other: CGM/CKM — Continuous Ketone Monitor will be applied at the start of Test Day 1. The sensor will be checked by the study team at each test day and will be removed and replaced by a fresh sensor at ~2- week intervals during the study. The sensor will be removed at the end of the final test day
Radiation: DXA — Lean Body Mass will be assessed once via DXA
  Arms: Control
Other: Urine Analysis — Prior to consumption of the Study Product, participants will be asked to completely void bladder. And hydration status will be determined via urine specific gravity (USG) reporting <1.025. Urine passed after the ingestion of the study product will be collected in a plastic container; participants will be asked to void their bladder and collect urine at the end of the test day. The volume produced will be recorded at the end of the study and aliquots will be frozen and stored for future analysis

SUMMARY:
One important difference between KE compounds is the ketone-promoting components, which determines the circulating ratio of blood ketone bodies, BHB and AcAc, and may in turn lead to important metabolic and signaling differences. Whereas some actions of the ketone bodies BHB and AcAc are shared, R-BHB has a broad range of signaling functions that are distinct from AcAc, some of which are shared by the non-circulating, non-oxidizable enantiomer, S-BHB. AcAc also has metabolic and signaling actions that are independent of BHB and is selectively oxidized in some cells that cannot oxidize BHB. Furthermore, responses to different ketone bodies vary between tissue types. A second difference between KE arises from the balance between direct delivery of ketones compared to indirectly elevating ketone concentration via metabolism of non-classical or classical ketogenic precursors. Classical ketogenesis itself may drive adaptation and some of the functional benefits associated with ketosis. BDO is included in all of the KE compounds, but it is currently unknown how consumption of BDO alone, and its metabolism via non-classical ketogenesis acutely affects metabolism. Additionally, ketogenesis is now understood to occur in certain cells outside the liver with important local biological effects, for example ketogenesis driven by medium chain fatty acids has been reported in astrocytes in vitro. Provision of systemic BHB by a KE may elicit different biological effects in some tissues such as the brain versus promoting in situ ketogenesis in that tissue. Overall, not only are functional effects of KE incompletely defined, but also it is unknown which effects are common to all KE versus which are specific to an individual KE compound (i.e., BHB Monoester vs AcAc Diester) or which may be attributable to the BDO precursor common to all of the KE. This study will be the first comparative full crossover study of all available KE and the precursor BDO at two serving sizes. Outcomes will focus on established effects of the BHB Monoester (including the effects on ketones, glucose and acid-base balance) and compare these with the effects of the AcAc Diester, C8 Ketonef Diester and BDO.

DETAILED DESCRIPTION:
BHB Monoester, C8 Diester, and (R) 1,3 Butanediol are commercially available in the products 'deltaG' (TdeltaS Global, FL, USA), 'Cognitive Switch' (Juvenescence Ltd, NJ, USA) and 'Avela' (Genomatica, CA, USA), respectively. The AcAc Diester is commercially available and is currently being used in clinical studies of Angelman's Disease. Therefore, we will standardize KE dosing to LBM (assessed using DXA) for all trials at 180 and 360 mg/kg LBM, which for a participant with 70 kg of lean mass corresponds to ~12.5 and 25 g, respectively. These doses are representative of typical commercial serving sizes and are expected to elevate blood BHB in the range of 1.5 - 2 mM39,61. All KEs will be consumed in their finished commercial form. As the KEs have different delivery matrices and flavorings (water-based beverage, emulsion beverage, gel capsules), we will not blind participants to each condition as this will not alter the metabolic outcomes of interest. Screening Visit: Participants that meet the initial qualifying criteria will visit the study center for a screening meeting in a private office to discuss the informed consent form with research team. The informed consent form will be provided to the participant for their review, the study will be described in full detail and any questions the interested participant has will be encouraged and responded to. The participant will be informed that even if they have signed the consent form, their participation in the study is dependent on anthropometric measures and diet and medical questionnaire answers to determine if they meet the study criteria. If the participant provides consent, they will be provided with questionnaires including Automated Self-administered 24-hour Dietary Assessment Tool (ASA24®),and medical history. All collected samples and data will be coded to maintain participant anonymity. We will give the participants a small volume of Study Product to screen for tolerance of the bitter tasting Study Products. We will also measure height, weight, BMI and body composition using a DXA scanner. If the participant is eligible for the study and is still interested in participating then they will be randomized to a study product order and scheduled to return to the study center for the first testing visit. Eligible participants will report to the study center in compliance with pre-test instructions (fasted > 10h, no alcohol >24h, no exercise >24h, consumed pre-test food). Upon testing day, participants will complete a baseline Beverage Tolerability Questionnaire (BTQ) and satiety visual analogue scale. Participants will be asked to completely void their bladder and a sample will be analyzed for hydration status. Bluetooth heart rate monitor chest strap will be administered. A study team member will assist the participant with application of a continuous ketone meter into the back of the arm, this will be removed and replaced with a fresh sensor at Test Days at ~2-week intervals; the sensor will be removed 24 hours after the cessation of the last in lab testing bout. Participants will be given written instructions on how to remove and dispose of monitor. A trained member of the study team will insert an IV cannula into a vein in the antecubital fossa to allow for repeated blood sampling. The cannula will be flushed with a small volume of saline after each sample withdrawal to maintain patency. We will collect 56mL of blood (7 x 8mL tubes) per testing day, which will be about 504mL of blood for the entire study. This is about 2.1 cups of blood. We will also collect capillary blood samples from a finger for real-time analysis of blood BHB and glucose concentration, using lancing device, commercially available test strips and a handheld monitor (KetoMojo, CA, USA). Participants will wear a fitted facemask connected to a metabolic cart for 10 minutes to collect measures of respiratory gas exchange. Participants will exhale once into a commercially available handheld breath acetone analyzer (Readout, MI, USA). Baseline blood sample, baseline respiratory gas measures and baseline breath acetone will be collected. Participants will then consume the Study Product that they were randomly allocated for that Test Day (details of Study Products attached in other files). Time of ingestion should be +/- 60 minutes from the time established at Test Day 1; they will be given 5 minutes to consume the Product. After Study Product consumption, they will remain at the study center for ~4 hours, repeating the aforementioned tests at 30min, 60 min, 90min, 180min & 240min. Participants will be asked to minimize ambulatory movement during the Test Day. Non caloric beverages (i.e.,water) will be permitted ad libitum and intake volumes will be recorded. At the end of each Test Day, the heart rate monitor and IV cannula will be removed and a dressing will be applied to the cannula site. Participants will be given a snack to consume before leaving the site.

ELIGIBILITY:
Inclusion Criteria:

* Male
* BMI between 18 and 29 kg/m2
* Aged 20 - 30 years
* Participant is willing and able to comply with all study procedures including the following prior to Test Days: fasting (>10 h; water only), no alcohol (>24 h), no exercise (>24 h), no acute illness and controlled feeding before each Test Day, maintain diet, exercise, medication, and supplement habits throughout the study.
* Participant has no health conditions that would prevent completion of the study requirements as judged by the Investigator based on health history.
* Participant understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Investigator.

Exclusion Criteria:

* Participant follows a low-carbohydrate diet (<30% energy from carbohydrate) or have used exogenous ketone supplements within 4-months of study participation.
* Participant has a Primary Care Physician diagnosed history or presence of uncontrolled and/or clinically important hypertension (blood pressure >150/95 mmHg), pulmonary, cardiac, hepatic, renal, endocrine (including type 1 and 2 diabetes), hematologic, immunologic, neurologic (e.g., Alzheimer's or Parkinson's diseases), psychiatric (including unstable depression and/or anxiety disorders) or biliary disorders.
* Participant has a known allergy, intolerance, or sensitivity to any of the ingredients in the study beverages, including soy and milk protein, wheat, shellfish, fin fish, eggs, tree nuts or peanuts (production facility handles nuts).
* Participant has unstable use of a medication or supplement that the Investigator considers may affect the outcomes of the trial.
* Consumption of alcohol more than 3 drinks per day or more than 18 drinks per week.
* Consumption of tobacco.
* Consumption of cannabis.
* Participant is currently in another research study or has been in the 14 days before screening.
* Participant has had a blood draw or donation in the last 8 weeks.
* Participant has a clinically important gastrointestinal (GI) condition that would potentially interfere with the evaluation of the study beverage [e.g., inflammatory bowel disease, irritable bowel syndrome, chronic constipation, severe constipation (in the opinion of the Investigator), history of frequent diarrhea, history of surgery for weight loss, gastroparesis, systemic disease that might affect gut motility according to the Investigator, medication managed reflux and/or clinically important lactose intolerance].
* Participant has a condition the Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the participant at undue risk.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study aims to recruit a homogenous, military relevant population to remove the confounding effects of variation in phenotype on exogenous ketone metabolism as far as possible. Thus, we will 15 recruit healthy and normally-active resistance/endurance trained men from the ages of 20-30 yr that represents typical active-duty military personnel.
Enrollment: 14 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Total Plasma Ketone AUC | Up to ~ 4 weeks
  Difference in total plasma ketone appearance (AUC) between the two serving sizes of study products and control

SECONDARY OUTCOMES:
Capillary d-BHB concentrations | Up to ~ 4 weeks
  Differences in ketone appearance during testing days
AcAc, R-BHB and S-BHB changes across trials | Up to ~ 4 weeks
  Differences in other blood ketones between the two serving sizes of study products and control. This will allow us to deduce specific ketone bodies during intervention.
Continuous Ketone and Glucose Monitoring | Up to ~ 4 weeks
  Diurnal concentrations of ketones and glucose via a continuous monitor. The ketone sensor in this CKM device is similar to the FreeStyle Libre continuous glucose monitoring (CGM). The sensor adheres to the back of the arm where it continuously samples interstitial fluid for quantification of BHB concentration. The sensor is worn for a period of 2-wk, three sensors will be used to cover all test days in this study (6 weeks). The first sensor will be inserted with assistance from the study team at the start of Testy Day 1, it will be checked every visit and replaced at Test Days following ~2-week intervals. The sensor will be removed 24 hours after the cessation of the last in lab testing bout (Testing Day 9). Participants will be given written instructions on how to remove and dispose of monitor. Feasibility, stability and other quality control parameters of this CKM/CGM has been established.
Ketone Excretion | Up to ~ 4 weeks
  Changes in urine excretion analysis
Ketone in breathe expiration | Up to ~ 4 weeks
  Concentration in breathe acetone via hand held reader
Alanine Change | Up to ~ 4 weeks
  Concentrations in blood metabolites will be determined using standard enzymatic assays.
Lactate Change | Up to ~ 4 weeks
  Concentrations in blood metabolites will be determined using standard enzymatic assays.
Free Fatty Acid Change | Up to ~ 4 weeks
  Concentrations in blood metabolites will be determined using standard enzymatic assays.
Heart Rate Variability | Up to ~ 4 weeks
  Changes in heart rate and heart rate variability
Satiety Visual Analogue Scale | Up to ~ 4 weeks
  We will use a 3-item visual analogue scale, that assesses hunger, fullness and desire to eat by participant's marking on a line anchored at either end with 'not at all' and 'extremely.' Distance along the line is measured in mm.
Beverage tolerability questionnaire (BTQ) | Up to ~ 4 weeks
  Ten tolerability issues are included in the BTQ: gas/flatulence, nausea, vomiting, abdominal cramping, stomach rumbling, burping, reflux (heartburn), diarrhea, headache, and dizziness. Participants are asked if the issue was present (pre- beverage - baseline) or had occurred since they took the study beverage (post-beverage - 4h) at the following intensities: none, mild (awareness of symptoms but easily tolerated), moderate (discomfort enough to interfere with but not prevent daily activity) or severe (unable to perform usual activity). These correspond to scores of 0-3, respectively for each issue, giving a maximal composite score, defined as the sum of the ten items, of 30.
Insulin | Up to ~ 4 weeks
  Differences in blood hormones insulin after supplementation will be analyzed using commercially available ELISA assay kits (Cayman Chemical, USA).
Ghrelin | Up to ~ 4 weeks
  Differences in blood hormones ghrelin after supplementation will be analyzed using commercially available ELISA assay kits (Cayman Chemical, USA).
Acid-Base Balance | Up to ~ 4 weeks
  Differences in blood acid-base balance (bicarbonate, strong ions)
Respiratory Gas Exchange | Up to ~ 4 weeks
  Differences in respiratory gas exchange (VO2 and VCO2)
Whole blood clinical chemistry | Up to ~ 4 weeks
  Whole blood clinical chemistry will be performed using a commercially available, clinical grade handheld analyzer (iSTAT, Abott, USA) and cartridges which will deliver the following data: Sodium, Potassium, pH, PCO2, Urea Nitrogen, Glucose, Hematocrit, TCO2, HCO3, Base Excess, Anion Gap, Hemoglobin (EC8+, Abott, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Jeff S Volek, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: OSU Office of Responsible Research Practices — https://orrp.osu.edu/

DOCUMENTS (2):
  • Study Protocol (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT05501366/Prot_000.pdf
  • Informed Consent Form (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT05501366/ICF_001.pdf